CLINICAL TRIAL: NCT04051047
Title: An Early Phase 1 Trial of Gemcitabine in Newly-Diagnosed Diffuse Midline Glioma
Brief Title: Gemcitabine in Newly-Diagnosed Diffuse Midline Glioma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Withdrawn by Principal Investigator
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UMCC 2018.159; HUM00135182 (Other: University of Michigan)
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Glial Tumor of Brain; Diffuse Intrinsic Pontine Glioma; Glioma
Keywords: Glioma
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Glioma | interventions — Gemcitabine; Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gemcitabine (Experimental): Gemcitabine will be given at 2100 mg/m2 IV over 30 minutes within 4 hours of planned surgical procedure. The surgical procedure is standard of care.
  Interventions: Drug: Gemcitabine; Procedure: Tumor biopsy and blood draw

INTERVENTIONS:
Drug: Gemcitabine — Participants receive a one time IV dose of gemcitabine prior to having standard of care surgery.
  Other Names: Gemzar
Procedure: Tumor biopsy and blood draw — As part of standard of care, all participants will undergo tumor biopsy and collection of peripheral blood.

SUMMARY:
The primary aim of this study is to determine the presence of gemcitabine in childhood diffuse midline gliomas (DMG) (previously classified as diffuse intrinsic pontine glioma [DIPG]) after systemic treatment with the drug.

DETAILED DESCRIPTION:
Participants in this study will be given a one-time, intravenous (IV) dose of gemcitabine prior to having standard-of-care surgery. During surgery, biopsies will be obtained for clinical and research purposes along with a blood sample. Cerebrospinal Fluid (CSF) is optional and will only be obtained if clinically indicated. This will be determined by the investigators and the provider performing the procedure.

Because patients will be undergoing a biopsy/resection as part of their standard-of-care therapy, this is an optimal time to obtain a tumor biopsy for this study. The biopsy will serve to see if the study drug is penetrating the tumor. Patients will then enter a follow-up period for 30 days post-surgery.

This trial is in conjunction with a University of Colorado trial started in 2016, "Gemcitabine in Children With Newly-Diagnosed Diffuse Intrinsic Pontine Glioma" (NCT02992015).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 3 years and less than 18 years at the time of enrollment.
* Patients must meet both of the first two conditions, OR the third:

  * Clinical findings consistent with a presumed new diagnosis of diffuse midline glioma (DMG) in the opinion of the treating neuro-oncologist, AND
  * Brain MRI findings consistent with a new diagnosis of DMG based on multidisciplinary consensus after review of imaging
  * OR, recurrent DMG requiring tumor resection or biopsy
* Adequate bone marrow, liver, renal and metabolic function (per protocol)
* Adequate coagulation defined as Prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ upper limit of normal (ULN ) for age
* Patients must meet one of the following performance scores:

  * ECOG performance status scores of 0, 1, or 2; 8
  * Karnofsky score of ≥ 60 for patients > 16 years of age; or
  * Lansky score of ≥ 60 for patients ≤ 16 years of age
* DMG biopsy/resection is planned for the clinical care of the patient independent of study participation by the treating pediatric neurosurgeon and neuro-oncologist.
* Informed consent and assent obtained as appropriate.

Exclusion Criteria:

* Pregnant or breastfeeding patients are not eligible due to teratogenic effects seen in animal/human studies
* Patients who have received any tumor-directed therapy prior to biopsy are not eligible. Concurrent treatment with corticosteroids is allowed.
* Any tumor-specific or clinical features that make surgical intervention unsafe in the opinion of the treating neurosurgeon.
* Patients with personal or family history of bleeding disorders are not eligible.
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements are not eligible.
* Patients with known hypersensitivity to gemcitabine

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-11-30 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with detectable intratumoral gemcitabine after systemic treatment with the drug | Day 1
  Gemcitabine will be considered to be detectable in a participant's tumor sample if gemcitabine or one of its metabolites (difluorodeoxyuridine [dFdU] or gemcitabine triphosphate [dFdCTP]) is detected at a measurable level in any of the participant's tumor samples. Undetectable gemcitabine will be defined as gemcitabine, dFdU, and dFdCTP levels below the detectable limits for all of an individual participant's samples, in the setting of detectable gemcitabine, dFdU, or dFdCTP in the plasma and/or cerebrospinal fluid (CSF) for that patient, and the pathologic review showing viable tumor tissue.

SECONDARY OUTCOMES:
Concentration of gemcitabine in patient tumor sample | Day 1
  Gemcitabine, dFdU and dFdCTP will be quantified in the available tumor sample(s), in plasma, and in CSF (if available). For this pilot trial, gemcitabine PK results will be analyzed descriptively, and this trial is not designed for statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Koschmann, M.D., Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No